CLINICAL TRIAL: NCT03510299
Title: Videoscope Guided Flexible LMA Insertion : Comparison With Blind Insertion
Brief Title: Videoscope Guided Flexible LMA Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-DEV-OBS-16-444
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Ideal Position of LMA Flexible

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Device: Control
- McGrath group (Experimental)
  Interventions: Device: Mcgrath

INTERVENTIONS:
Device: Mcgrath — McGrath assisted insertion of LMA flexible
  Arms: McGrath group
Device: Control — Digital manipulation technique of LMA flexible insertion
  Arms: Control group

SUMMARY:
Laryngeal Mask Airway Flexible (LMA Flexible) is useful in various surgery because of its unique design. The flexometallic tube allows it could be used in head and neck related surgery but also make insertion more difficult. The ideal position of LMA Flexible is important because in most case, the surgery requiring LMA Flexible allows movements of the stem or patient's head during operation without dislodgement of LMA Flexible. Several studies have examined different techniques like assisting LMA Flexible with rigid introducers or lifting epiglottis with direct laryngoscope. But there is no study using videolaryngoscope (VL) for LMA Flexible insertion. The investigator hypothesized that McGrath(McGRATH™ MAC video laryngoscope;Aircraft Medical Ltd, UK.), one kind of the VL, assisted insertion would increase the success rate of LMA Flexible insertion by lifting epiglottis and securing a view while LMA Flexible is seated. The aim of this study was to investigate the efficacy of the McGrath VL assisted insertion of LMA Flexible compared with the standard method of digital manipulation technique in regard to the ideal anatomical position and sealing pressure in anesthetized adult patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American society of anesthesiologist) physical status classification system I and II,
* scheduled to elective general anesthesia with the use of LMA

Exclusion Criteria:

* suspected difficult airway
* a history of a recent upper airway tract infection
* gastroesophageal reflux
* body mass index > 30 kg/m2

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Ideal positioning rate of LMA flexible | 3 minute after LMA flexible insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Jiyoung Yoo, Suweon, Kyunggido, South Korea

IPD SHARING:
Plan to Share IPD: No